CLINICAL TRIAL: NCT01827696
Title: Effect of American Ginseng on Exercise-induced Muscle Soreness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Peter Lemon, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Muscle Damage
Keywords: Muscle; Soreness; Muscle function; Damage; Ginseng
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): American Ginseng ingestion
  Interventions: Dietary Supplement: Ginseng
- Placeobo (Placebo Comparator): non-active ingredient
  Interventions: Dietary Supplement: Ginseng

INTERVENTIONS:
Dietary Supplement: Ginseng — Effect of four weeks of daily Ginseng intake (2gm/day) on muscle soreness following downhill running exercise

SUMMARY:
Healthy participants will ingest American ginseng daily or a placebo for four weeks prior to engaging in a unaccustomed exercise bout designed to induce mild-moderate muscle soreness. Muscle soreness will be assessed via decrements in muscle strength and with a self-rating of perceived soreness before and several times after the exercise.

DETAILED DESCRIPTION:
Healthy men and women will consume either 2000 mg of American ginseng daily (four 500 mg pills will be taken at four different times during the day always with food/meals) or a placebo (4 cellulose) for four weeks prior to engaging in a 40 minute downhill treadmill jog (12% decline) at a speed of 7 miles per hour. Participants will consume one pill with breakfast, one pill with lunch, one pill with dinner and another pill with a snack either between meals or prior to bedtime. The exercise will be consist of five, eight minute bouts of jogging with two minutes of rest/recovery in between. The degree of muscle soreness will be assessed using a Biodex strength testing machine (isometric and concentric isokinetic torque), and a self-rating of perceived soreness on a scale from zero to ten. All of the above measures will be taken before and several times after the downhill jogging protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women, (women must weigh between 55-65 kg., while men must weigh between 75-85kg).
* Participants must not have engaged in any endurance run training in the past 9 months.

Exclusion Criteria:

* Injured
* Regular runners
* Pregnant (or with any chance they may become pregnant)
* Breast-feeding
* Diabetics or those taking medication for diabetes
* Insomniacs
* Schizophrenics
* Hyper- or hypotension
* Cancer
* Irregular heartbeats
* Heart disease
* Females with endometriosis or uterine fibroids
* Those who have surgery scheduled during the study or within the two weeks following the completion of the study
* Those taking warfarin or medication for depression.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
muscle strength | 1 month
  ginseng & muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Peter WR Lemon, PhD, Principal Investigator — Western University, Canada
Locations (1):
- University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung HL, Kwak HE, Kim SS, Kim YC, Lee CD, Byurn HK, Kang HY. Effects of Panax ginseng supplementation on muscle damage and inflammation after uphill treadmill running in humans. Am J Chin Med. 2011;39(3):441-50. doi: 10.1142/S0192415X11008944. PMID 21598413